CLINICAL TRIAL: NCT04728165
Title: Pilot Study to Explore the Anti-Inflammatory Effects of Time-Restricted Feeding
Brief Title: Anti-Inflammatory Effects of Time-Restricted Feeding
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 10000149; 000149-H
Record Dates: First submitted 2021-01-27; First posted 2021-01-28 (Actual); Last update posted 2025-06-12 (Actual); Status verified 2025-06-10

CONDITIONS: Psoriasis; Systemic Inflammation
Keywords: Psoriasis; GLUCOSE METABOLISM; insulin metabolism; NLRP3 Inflammasome; Th17 inflammation; Natural History
MeSH Terms: conditions — Psoriasis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- control group: Age (+/-5 yrs) and BMI (+/- 5 kg/m2) matched control male subjects for inclusion in the control group
- psoriasis group: Males between the ages of 18 and 70 with mild to moderate active psoriasis by PASI score for inclusion in psoriasis group

SUMMARY:
Background:

Time-restricted feeding (TRF) means that a person eats only during certain hours of the day. In other studies, researchers have found that fasting can improve immune system function in healthy people. They want to see if TRF has the same effect on people with psoriasis.

Objective:

To test whether TRF can change metabolism and decrease some markers of inflammation in the blood of people with mild to moderate psoriasis.

Eligibility:

Males ages 18 to 80 with mild to moderate active psoriasis, and healthy volunteers

Design:

Participants will be screened with a medical history and medicine review. They will have a physical exam and blood tests. Their skin will be examined. They will have a nutritional evaluation. Their resting energy expenditure will be measured. For this, a clear plastic ventilation hood will be placed over the head for a short time.

Participants will stay at the NIH Clinical Center for 4 1/2 days. They can watch TV, do work, do schoolwork, and other quiet activities.

A small sensor will be placed under participants skin to measure blood glucose.

For part of the study, participants will be housed in a small room called a metabolic chamber. They will wear a heart monitor.

Participants will walk on a treadmill for 30 minutes each day at a comfortable speed.

For 3 days, participants will eat all their daily calories between 8 am and 2 pm. They will fast for the other 18 hours of the day. They can drink water.

Participants will complete mixed meal tests. They will drink a liquid meal for breakfast. Then they will give blood samples via intravenous (IV) catheter.

Participation will last for 5 days....

DETAILED DESCRIPTION:
Study Description:

Fasting and caloric restriction interventions have anti-inflammatory effects, although the underling regulatory controls are poorly characterized. This pilot study will explore transcriptional profiles in various leukocyte populations comparing the effect of time restricted feeding (TRF - 6-Hr feeding/18-Hr fast) to a more conventional dietary regimen (12-Hr feeding/12Hr fast). These regulatory effects will be evaluated in an inflammatory disease (psoriasis) in response to TRF and by comparing the relative response comparing the psoriasis population to a matched TRF control group.

Objectives:

1. Evaluate the effect of TRF on Th17 immunological signatures.
2. Compare the role of TRF on chromatin remodeling on CD4+ T cells, monocytes and neutrophils comparing control and

   psoriatic subjects.
3. Evaluate the effect of TRF on glucose and insulin metabolism and overall metabolic flexibility.

Endpoints:

The primary outcome will be the change in the secretion of IL-17 from activated CD4+ T cells from baseline to the end of TRF as a measure of biological reprograming in the psoriasis group and to assess the change in IL-17 release comparing the effects of TRF in the control versus psoriasis groups.

Secondary outcomes are:

1. Evaluate the effect of TRF on chromatin signatures of gene activation (ATACseq) and gene silencing (H3K9me3).
2. Explore the effect of TRF on low-density granulocytes, neutrophils and monocytes.
3. Evaluate whether TRF improves 24-hour glucose levels, glycemic excursions during a meal test and modulate sleeping

and feeding metabolic flexibility as defined by the change in sleeping respiratory exchange ratio from the daytime. (24-hr

substrate oxidation as defined by the averaged RER)

ELIGIBILITY:
* INCLUSION CRITERIA:

Individuals must meet the inclusion criteria listed below in order to be eligible to participate in the study.

* Males between the ages of 18 and 80 with mild to moderate active psoriasis by PASI score for inclusion in psoriasis group
* Age (plus or minus 10 yrs) and BMI (plus or minus 5 kg/m^2) matched control male subjects for inclusion in the control group.
* Ability to provide informed consent
* Willingness and ability to participate in study procedures

EXCLUSION CRITERIA:

* Severe psoriasis by PASI (Psoriasis Area and Severity Index) score > 12
* Treatment with systemic biologic immune modifying agents within the last 2 months.
* Currently on treatment for allergies or other inflammatory diseases.
* Has taken Vitamin B or tryptophan supplementation within 2 weeks of participation.
* Unwillingness/inability to provide informed consent.
* Individuals with known history of type 1 and 2 diabetes mellitus or other metabolic conditions that would interfere with study parameters including chronic kidney disease, chronic liver disease, history of hypoglycemia
* On treatment with medication that would interfere with study parameters including anti-hyperglycemic medications, systemic steroids, adrenergic-stimulating agents, other medications known to affect sleep, circadian rhythms or metabolism.
* Caffeine in excess of three 8 oz cups per day.
* Factors that affect circadian rhythm including individuals who perform overnight shift work, irregular sleep and/ or eating schedules, regularly fast for more than 15 hours/ day
* Regular use of tobacco product within last 3 months.
* Consuming more than 3 servings of alcohol/ day
* Engaged in competitive sports training
* Moderate to severe claustrophobia
* Unstable weight with more than 5% body weight change in last 3 months
* Food allergies or intolerances or dietary patterns that would prohibit consumption of the metabolic diet or mixed meal test.

Ages: 18 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Males between the ages of 18 and 70 with mild to moderate active psoriasis by PASI score for inclusion in psoriasis group Age (plus or minus 5 yrs) and BMI (plus or minus 5 kg/m2) matched control male subjects for inclusion in the control group. Ability to provide informed consent Willingness and ability to participate in study procedures
Sampling Method: Non-Probability Sample
Enrollment: 27 (Actual)
Dates: Start 2021-06-09 (Actual); Primary Completion 2023-07-28 (Actual); Study Completion 2023-07-28 (Actual)

PRIMARY OUTCOMES:
change in the secretion of IL-17 from activated CD4+ T cells from baseline to the end of TRF | 3 years
  The primary outcome will be the change in the secretion of IL-17 from activated CD4+ T cells from baseline to the end of TRF as a measure of biological reprograming in the psoriasis group and to assess the change in IL-17 release comparing the effects of TRF in the control versus psoriasis groups.

SECONDARY OUTCOMES:
Evaluate the effect of TRF on chromatin signatures of gene activation (ATACseq) and gene silencing (H3K9me3) | 5 years
  Evaluate the effect of TRF on chromatin signatures of gene activation (ATACseq) and gene silencing (H3K9me3)
Explore the effect of TRF on low-density granulocytes, neutrophils and monocytes | 5 years
  Explore the effect of TRF on low-density granulocytes, neutrophils and monocytes.
Evaluate whether TRF improves 24-hour glucose levels, glycemic excursions during a meal test and modulate sleeping and feeding metabolic flexibility as defined by the change in sleeping respiratory exchange ratio from the daytime. (24-hr substra... | 4 years
  Evaluate whether TRF improves 24-hour glucose levels, glycemic excursions during a meal test and modulate sleeping and feeding metabolic flexibility as defined by the change in sleeping respiratory exchange ratio from the daytime. (24-hr substrate oxidation as defined by the averaged RER)

CONTACTS AND LOCATIONS:
Overall Officials: Michael N Sack, M.D., Principal Investigator — National Heart, Lung, and Blood Institute (NHLBI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

REFERENCES:
- [Derived] Romero Arocha S, Han K, Huffstutler RD, Thota GP, Macheret NA, Courville AB, Brychta RJ, Chen KY, Chung ST, Coates LC, Clarke AJ, Sack MN. Effects of Acute Time-Restricted Eating on Inflammation in Individuals With Psoriasis: Protocol for a Case-Control, Prospective Study. JMIR Res Protoc. 2025 Aug 15;14:e74999. doi: 10.2196/74999. PMID 40815832
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_000149-H.html